CLINICAL TRIAL: NCT02644616
Title: The Safety and Efficacy of Tolvaptan for Patients With Tricuspid Regurgitation and Right Heart Failure After Left Heart Valves Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Yuan Fang, Principal Investigator, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156-ZOC-1401
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Tricuspid Regurgitation; Right Heart Failure
Keywords: tolvaptan; safety and efficacy; left heart valves replacement
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trial group(tolvaptan group) (Active Comparator): trial group (tolvaptan 15mg/d po(10 days) + torasemide 20mg/d iv,n=20)
  Interventions: Drug: tolvaptan+torasemide
- control group (Placebo Comparator): control group(placebo 15mg/d po(10 days) +torasemide 20mg/d iv,n=20)
  Interventions: Drug: placebo+torasemide

INTERVENTIONS:
Drug: tolvaptan+torasemide — tolvaptan 15mg/d po(10 days) + torasemide 20mg/d iv
  Arms: trial group(tolvaptan group)
Drug: placebo+torasemide — placebo 15mg/d po(10 days) +torasemide 20mg/d iv
  Arms: control group

SUMMARY:
The investigators research the early improvement of fluid retention and mid-term prognosis through the administration of tolvaptan for the patient with tricuspid regurgitation and right heart failure after left heart valves replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with tricuspid regurgitation and right heart failure after left heart valves replacement
2. Patients who takes existing diuretic
3. The patient is willing to participate in the study

Exclusion Criteria:

1. Patients with hypersensitivity to study drug
2. Anuric patients
3. Patients with hypernatremia
4. Female patients who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant
5. Malignant tumor
6. Patients with serious hepatic disorder or Serious Renal failure
7. Patients otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The change of all the subjects'liquid intake and output volume change after a period(10 days) of treatment | 2015.01-2017.12

SECONDARY OUTCOMES:
A cumulative urine volume for 72 hours (all subjects) | 2015.01-2017.12
Echocardiography results VS the baseline results(all subjects) | 2015.01-2017.12
Change of right heart failure signs(all subjects) | 2015.01-2017.12
Onset of cardiovascular event (all subjects) | 2015.01-2017.12
Onset of serious adverse event(all subjects) | 2015.01-2017.12
other adverse events(all subjects) | 2015.01-2017.12

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yuan, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- FangYuan, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan F, Wu Z, Jiang L, Zhou J, Xu L, Liu H, Ma L, Zhai Z, Zhang J. Short-Term Effects of Tolvaptan in Tricuspid Insufficiency Combined with Left Heart Valve Replacement-Caused Volume-Overload Patients: Results of a Prospective Pilot Study. Am J Cardiovasc Drugs. 2019 Apr;19(2):211-218. doi: 10.1007/s40256-018-0304-1. PMID 30255476